CLINICAL TRIAL: NCT04630080
Title: Scalp Cooling Study for the Prevention of Chemotherapy-induced Alopecia in Chinese Breast Cancer Patients
Brief Title: Alopecia Prevention Scalp Cooling in Chinese Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Yeo, Professor, Department of Clinical Oncology, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SYM013
Record Dates: First submitted 2020-10-21; First posted 2020-11-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scalp Cooling (Experimental)
  Interventions: Device: Scalp cooling

INTERVENTIONS:
Device: Scalp cooling — Scalp cooling is a physical method to reduce chemotherapy-induced alopecia

SUMMARY:
The Orbis Paxman Hair Loss Prevention System is a new equipment introduced to Hong Kong in 2017. Although this device has been widely used in the United States, Europe and Australia, acceptability, efficacy and safety data in Chinese have not yet been available. The objective of this prospective study is to collect clinical data in Chinese patients using the Orbis Paxman Hair Loss Prevention System to prevent chemotherapy-induced alopecia.

This project seeks to demonstrate that the Orbis Paxman Hair Loss Prevention System is safe and effective in reducing chemotherapy-induced alopecia in woman with breast cancer undergoing neoadjuvant or adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

i) New diagnosis of breast cancer stage I-III

ii) Chinese ethnicity

iii) ECOG 0-1

iii) Planning to undergo neoadjuvant or adjuvant chemotherapy with curative intent

iv) Chemotherapy must be planned for at least 4 cycles of full-dose anthracycline and/or taxane based chemotherapy regimen,

1. Defined as one of the following regimens:

   * Adriamycin 60 mg/m2 with cyclophosphamide 600 mg/m2 for 4 cycles (AC) > 5-Fluorouracil 500 mg/m2, Epirubicin 100mg/m2, and cyclophosphamide 500 mg/m2 for 3 cycles, followed by Docetaxel 100 mg/m2 for 3 cycles (FEC-D)
   * AC x 4 cycles, followed by Docetaxel 100 mg/m2 for 4 cycles (AC-D)
   * AC x 4 cycles, followed by Paclitaxel 175 mg/m2 for 4 cycles (AC-P)
   * Docetaxel 75 mg/m2 with cyclophosphamide 600 mg/m2 for 4-6 cycles (DC)
   * Docetaxel 75 mg/m2 with carboplatin AUC of 5-6 for 4-6 cycles (DCb)
2. Concurrent trastuzumab and/or pertuzumab at standard doses is allowed.
3. Administration of chemotherapy on a dose dense schedule with GCSF is allowed.

v) Adequate organ functions vi) Normal thyroid stimulating hormone vii) Subjects with history of diabetes must have acceptable HBA1c on study entry viii) Subjects who provide consent and are mentally competent and able to fill in study questionnaires

Exclusion Criteria:

i) Subjects with any other concurrent malignancy including hematological malignancies (i.e. leukemia or lymphoma)

ii) Subjects with cold agglutinin disease or cold urticaria

iii) Age ≥ 70 years

iv) Personal history of migraines, cluster or tension headaches as defined as actual medical diagnosis by a physician and/ or prescribed medications. If personal history of migraines was related to a past medical problem that is now resolved, subject may go on study at the discretion of the Principal Investigator.

v) Elevated liver enzymes or bilirubin defined as 3 times the upper limits of normal

vi) Serum Albumin < 3.0

vii) Subjects with anemia (defined as a hemoglobin < 10)

viii) Subjects who have lichen planus or lupus, or other dermatological conditions involving scalp

ix) Subjects who are underweight (defined as a BMI < 18.5)

x) Subjects who have had previous chemotherapy exposure

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of scalp cooling in preventing chemotherapy-induced alopecia | 2 year

SECONDARY OUTCOMES:
The rate of preceived hair preservation during and after completion of chemotherapy | 2 years
  It will be assessed by study tool ALOPECIA ASSESSMENT BY PATIENT AND WIG USE FORM
The quality of life during and after completion of chemotherapy | 2 years
  It will be assessed by study tool EORTC QLQ-30
The disease site specific quality of life during and after completion of chemotherapy | 2 years
  It will be assessed by study tool EORTC QLQ - BR23
The incidence of treatment-emergent adverse events of scalp cooling | 2 years
  It will be assessed by COMFORT SCALE FORM.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, MD, FRCP, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hosptial
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No